CLINICAL TRIAL: NCT06264895
Title: Evaluation of a Low-threshold Exercise And Protein Supplementation Intervention for Women (LEAP-W) Experiencing Homelessness and Addiction: Protocol for a Single Site Intervention Study.
Brief Title: Protocol for a Low Threshold Exercise Intervention for Women Experiencing Homelessness and Addiction.
Acronym: LEAP-W
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Julie Broderick, Dr. Julie Broderick, Assistant Professor, Head of Discipline of Physiotherapy, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trinity College Dublin 211202
Record Dates: First submitted 2024-02-06; First posted 2024-02-20 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Social Exclusion; Chronic Disease; Physical Disability; Addiction
MeSH Terms: conditions — Social Isolation; Chronic Disease; Behavior, Addictive | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: single -arm longitudinal cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of an exercise intervention for women experiencing homelessness and addiction. (Experimental): A 3 times weekly exercise intervention with protein supplementation will be delivered to all study participants for 10 weeks.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — three times weekly exercise intervention with protein supplementation

SUMMARY:
Background: Frailty is a complex multi-dimensional state of increased vulnerability to adverse health outcomes and is usually associated with older age but there is growing evidence of accelerated ageing and frailty in non-geriatric populations, including those experiencing socio-economic deprivation and extreme social exclusion, such as people experiencing homelessness. Addiction, as a coping mechanism for prior trauma, is common among people who are homeless and can have a gendered dimension. Women experiencing homelessness and addiction have unique needs which require a gendered approach. The aim of this study is to explore the effectiveness of an exercise intervention to target the known physical functioning deficits and frailty which this population experiences.

Methods: This mixed-methods study will explore physical functioning deficits and frailty in women experiencing homelessness and addiction, using a bespoke test battery and an exercise intervention. Physical function (10m Walk Test, 2 Minute Walk Test, Single Leg Stance Test, Chair Stand Test, hand grip dynamometry), frailty (Clinical Frailty Scale and the SHARE-FI) and nutritional status (Mini-Nutritional Status), pain (Numerical Pain Rating Scale) and quality of life (SF 12-V2) will be evaluated. The intervention will involve a 3-times weekly exercise programme with protein supplementation for 10 weeks. Following this, qualitative interviews, which will be thematically analysed using Braun & Clarke methodology, will be conducted. This study will be conducted in Dublin from February to July 2024.

Discussion: Little is kn own about frailty-focussed interventions in women experiencing homelessness and addiction. This proposed study will help to increase the knowledge base regarding the physical health burden and frailty experienced by this extremely vulnerable population and will deliver a targeted intervention with a gendered dimension to mitigate its affects. The findings of this research will help narrow this research gap and will guide clinicians and policy makers to implement unique gender-based treatment strategies for this population.

DETAILED DESCRIPTION:
Previous linked research of exercise interventions in people experiencing homelessness, demonstrated high retention with excellent engagement and feedback from its female participants, yet caution was observed around engaging in a mixed exercised programme with men. Women have traditionally been underserved in research and policy, yet multiple sources cite women as the fastest growing homeless demographic. No study has examined how targeted women-only exercise programmes with nutritional supplementation work in practice in this population.

The overall aim of this study is to explore physical functioning and frailty outcomes of an exercise intervention with protein supplementation in a group of (non-geriatric) women experiencing homelessness and addiction challenges.

The objectives are:

1. To evaluate recruitment, retention and adherence rates, and any adverse effects of the intervention.
2. To evaluate pre- and post-intervention levels of physical, nutritional and frailty status, pain and general health status.
3. To evaluate programme feedback and gain deeper insights into participants perspectives and experiences of the exercise intervention.

This mixed-methods study will involve a single-arm intervention which will take place in Dublin city centre, in a day-service centre which provides services for women who are homeless and/or in addiction. Following the intervention qualitative research in the form of individual exit interviews will be conducted with 20 participants or up to the point of data saturation.

The 10-week intervention will involve a low threshold, three-times weekly exercise programme (two exercise classes with protein supplementation and an outdoor 'Park Walk') delivered over 12 weeks to offer flexibility to participants. It will be delivered by two research physiotherapists who will adhere to all safety procedures. Further flexibility will be facilitated with the provision of a four-week window for pre-intervention evaluations prior to commencement of the programme, and group or one-to one sessions will be delivered based on participant preference. The exercise classes will be multi-modal, with a primary focus on strength and based on core set of resistance exercises. Aerobic, balance and flexibility work will be integrated into the class and the exercises will be individualised based on initial assessment results and presentation of participants. Using a gender-based perspective, the following considerations and adaptions will be built into the class; (i) core-stability exercises to target pelvic floor and/or abdominal muscle weakness, (ii) bone building exercises to target peri-and postmenopausal bone loss and (iii) age-associated muscle mass loss. Music, dance and fun orientated physical activity games, an important feature of prior linked studies, will be incorporated to optimize enjoyment and self-esteem. Borg's Rate of Perceived Exertion Scale will be used to monitor effort and scale the intensity of the workout. To promote post-exercise muscle protein synthesis, a nutritional supplement (200ml pre-prepared 'protein shake', Fresubin) which consists of 20g of protein will be offered immediately post exercise. The 'Park Walk' will focus on the aerobic component of the intervention, using green open space to maximise physical and mental health outcomes. It will be a flexibly arranged 20-30 minute self-paced group or one-to-one walk. To build sustainability beyond the ten week programme brief health promoting and physical activity educational interventions will be included in the exercise class setting to empower people to engage in unsupervised exercise following the study. Following the intervention one-to-one in-person exit interviews will be conducted to enable participants to provide feedback and express personal views, in order to enhance the understanding of behaviours, adherence and retention challenges and to provide insights for future programmes in this area. Interviews will continue until 20 participants are seen or until data saturation is reached. The interviews will be audio-recorded and transcribed verbatim and member checking will be utilised.

Analytic plan: For quantitative data, nominal or ordinal variables will be reported as frequencies and percentages. Continuous variables will be summarised as mean and standard deviation if normally distributed and median and inter-quartile range if non-normally distributed. Data will be tested for normality using the Kolmogorov-Smirnov/Shapiro Wilk test and will be compared across timepoints using the general linear model procedure (normally distributed data) and the Friedman's test (non-normally distributed data). Chi-squared t-tests will be used where appropriate and some data may be categorised to investigate relationships between variables. Exploratory regression models will be developed to explore correlates and predictors of frailty and poor physical functioning. A p-value of <0.05 will be considered significant. For the qualitative data, Braun and Clarke thematic analysis methodology will be employed to provide an in-depth analysis of the exit interview data.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (18-65 years) accessing services in Jane's Place who consent to participation.

Exclusion Criteria:

* Any person not meeting the age eligibility criteria.
* Any person identifying as a male.
* Any person lacking capacity to give consent.
* Any person with major physical/medical or cognitive challenges which would preclude ability to safely complete the assessment or
* Any person with insufficient English language ability to give fully informed consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — any person identifying as female
Enrollment: 45 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 12 weeks
  Number recruited to the study
Retention | 12 weeks
  Number of repeat visits
Adverse events | 12 weeks
  An unfavourable and unintended sign, symptom or disease having been absent at baseline, or, if present at baseline, appears to worsen and is temporally associated with medical treatment or procedure, regardless of the attribution.

SECONDARY OUTCOMES:
Hand grip dynamometry | up to 10 weeks
  Strength will be measured using a hand-grip dynamometer
Limb circumference | up to 10 weeks
  Measurement of muscular mass at mid arm and mid calf circumference will be recorded.
10 Metre Walk Test | up to 10 weeks
  This test measures walking speed and functional mobility and is recorded in m/s. Gait speed is calculated as total distance/time.
2 Minute Walk Test | up to 10 weeks
  This test of self-paced walking ability and functional capacity assesses a participants' ability to walk unaided over a 15m distance, as fast as possible, for two minutes. Rest breaks are permitted and the distance covered is measured.
The Chair Stand Test | up to 10 weeks
  This tests lower limb strength and endurance and records the total number of sit to stand repetitions performed in 30 seconds.
Single Leg Stance Test | up to 10 weeks
  This balance test is performed on each leg. The participant is timed standing unassisted on one leg, with eyes open and hands placed on the hips.
Numerical Rating Scale (NRS) | up to 10 weeks
  The NRS is a unidimensional measure of pain intensity from 0-10, with 0 being zero pain and 10 the worst pain imaginable.
Clinical Frailty Scale (CFS) | up to 10 weeks
  The CFS is validated for people over 65 years. It is assessed by the tester. Each point on the scale correlates with a level of frailty and a visual chart aids the tester in classifying frailty from 1 (very fit) to 9 (terminally ill). Higher scores indicate higher levels of frailty.
SHARE-Frailty Instrument (FI) | up to 10 weeks
  The SHARE-FI consists of four brief questions related to the following variables; exhaustion, loss of appetite, walking difficulties and low physical activity. Grip strength will also be measured, and the five results are entered into a freely available web calculator to generate a frailty score and a frailty category of non-frail, pre-frail and frail is generated.
Mini Nutritional Assessment (MNA) | up to 10 weeks
  The MNA assesses the risk of malnutrition. It consists of six questions on food intake, weight loss, mobility, psychological stress, or acute disease, the presence of dementia or depression, and body mass index (BMI). The maximum is 14. A score of 12-14 indicates normal nutritional status and a score of 7 or less indicates malnourishment.
Short Form-12 V2 | up to 10 weeks
  The SF-12 V2 is a self-report measure of health. It uses eight domains including physical and social activities, pain, mental health, emotional health, vitality and general health perceptions to measure health. The tester will read and complete the 12-question survey with the participant. Results will be entered into a software program provided by the licensing company QualityMetric and two summary scores, mental health (MCS12) and physical health (PCS12) will be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Broderick, PhD, Principal Investigator — Trinity College, University of Dublin, Dublin, Ireland
Locations (1):
- Trinity College Dublin, University of Dublin, Dublin, Ireland

REFERENCES:
- [Derived] Kennedy F, Murray D, Ni Cheallaigh C, Romero-Ortuno R, Gavin S, Broderick J. Exploring the impact of targeted exercise in women experiencing homelessness, addiction and mental health challenges: a mixed-methods feasibility study. BMJ Open. 2026 Feb 6;16(2):e103060. doi: 10.1136/bmjopen-2025-103060. PMID 41651532